CLINICAL TRIAL: NCT04476329
Title: A Randomized Phase II Study of First Cycle Optimization for Regorafenib Treatment Compared to Standard Dose of Regorafenib in Patients With HCC Who Failed Any 1st Line Systemic Treatment and for Whom the Physician is Intending to Treat With Regorafenib
Brief Title: Optimization for Regorafenib in HCC
Acronym: ReDos HCC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment rate not sufficient to meet funding entity's corporation timeline expectations, entity terminated study's fiscal support. Termination decision was purely administrative in nature and did not involve drug or patient safety issues.
Sponsor: SC Liver Research Consortium, LLC (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21305
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Liver Cancer; HCC; Regorafenib; Sorafenib; Stivarga
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — regorafenib

STUDY DESIGN:
Intervention Model Description: Arm A will initiate Cycle 1 treatment at 80mg daily of regorafenib escalating up to but not exceeding 160mg daily at 40mg per week increments.
  Arm B will initiate Cycle 1 treatment at 160mg daily of regorafenib.
Masking Description: This trial will not be masked, subjects will know which arm they are randomly assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Active Comparator): Arm A: Regorafenib Cycle 1:
  * 80 mg daily Week 1
  * 120 mg daily Week 2
  * 160 mg daily week 3 then 1 week off followed by Cycle 2+ (160 mg for 21 days/1 week off) Subsequent Treatment Cycles
  * 160 mg daily for 21 days, then 1 week off.
  Interventions: Drug: Regorafenib 40 MG
- B (Active Comparator): Arm B: Regorafenib Cycle 1:
  * 160 mg daily for 21 days/then 1 week off Subsequent Treatment Cycles
  * 160 mg daily for 21 days, then 1 week off
  Interventions: Drug: Regorafenib 40 MG

INTERVENTIONS:
Drug: Regorafenib 40 MG — Regorafenib (BAY 73-4506) is an oral small molecule tyrosine kinase inhibitor (TKI) that potently blocks multiple protein kinases, including kinases involved in tumor angiogenesis (vascular endothelial growth factor receptor [VEGFR] 1, 2, 3, Tyrosine kinase with immunoglobulin-like and epidermal growth factor-like domains 2 [TIE2]), stem cell growth factor receptor (KIT, rearranged during transfection [RET], p38-alpha, a member of the mitogen activated protein kinase [MAPK] family, proto-oncogene c-RAF [c-RAF], proto-oncogene BRAF [BRAF], BRAFV600E), metastasis (VEGFR3, platelet-derived growth factor receptor [PDGFR], fibroblast growth factor receptor1 [FGFR1]) and tumor immunity (colony stimulating factor 1 receptor [CSF1R]).
  Other Names: Stivarga

SUMMARY:
This is a randomized, two arm, phase II study of 1st Cycle dose optimization for regorafenib treatment compared to standard dose of regorafenib treatment in HCC patients for whom the physician is intending to treat with regorafenib and who failed any 1st line systemic treatment.

DETAILED DESCRIPTION:
In this study, the investigators intend to evaluate the regorafenib ReDOS strategy to optimize the dose of regorafenib in patients with unresectable HCC (uHCC) who progressed during or after the first-line systemic treatment. This would allow improving the tolerability profile for patients such as those not selected based on prior sorafenib tolerability. The proposed regorafenib dosing escalation strategy for subjects randomized to the Arm A starting 80 mg/day dose for one week (Cycle 1, Week 1) is, if absent significant drug-related toxicities, to escalate to 120 mg/day for another week (Cycle 1, Week 2), and then, again if absent significant related toxicities, escalate to a total dose of 160 mg/day (Cycle 1, Week 3) followed by a week-long break (Cycle 1, Week 4).

Arm B, the comparative arm, will include a standard dose/schedule regorafenib of a 160 mg/day starting on Cycle 1, Day 1. The primary goal of this Arm is compare whether, or not, an 80 mg/day starting dose of regorafenib that escalates weekly by 40 mg until 160 mg/day is non-inferior to the FDA approved labeling 160 mg starting dose of regorafenib in terms of Overall Survival (OS) in HCC subjects. The investigators will also compare the proportions of patients in each arm who complete two cycles of treatment and who intend to continue to a third cycle if no tumor progression is noted on the 8-week disease scan. Other outcomes such as Quality of Life measures, and toxicity profile with a focus on regorafenib related toxicities such as hand-foot skin reaction will also be assessed.

Patients will be randomized 1:1 to either Arm A receiving the Cycle 1 Week-1 80 mg daily dose or Arm B the standard FDA labeling 160 mg daily starting dose, with subsequent dose adjustments as needed. Patients with unacceptable toxicities at the 80 mg dose may be considered for further dose reduction but will no longer be included in the overall survival analysis. After the conclusion of Cycle 2 (Week 8 of treatment), if toxicities have sufficiently resolved, re-escalation is allowed 40 mg at a time every four weeks to a maximum of 160 mg/day at the discretion of the treating investigator.

Patients will continue treatment until progression, unacceptable adverse events, or patient refusal. Treatment will then be discontinued, and the patient will go to event monitoring.

Additionally, a site-optional and subject-optional sub-study collecting blood serum samples at the Screening Visit for "hold and store" for future analysis of CD14, CD15, and CD16 cells as well as other potential biomarkers to be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age ≥ 18 years.
2. Histological, cytological confirmation of hepatocellular carcinoma or non-invasive diagnosis of HCC as per American Association for the Study of Liver Diseases (AASLD) criteria in patients with a confirmed diagnosis of cirrhosis.
3. Locally advanced or metastatic and/or unresectable HCC that is not amenable or progressed after curative surgical and/or locoregional therapies.
4. Patients who received one prior systemic treatment and for whom the treating physician has decided to treat with regorafenib.
5. Life expectancy of ≥ 3 months.
6. The following laboratory values obtained ≤ 7 days prior to randomization.

   * Absolute neutrophil count (ANC) > 1500/mm3
   * Platelet count > 60,000/mm3
   * Hemoglobin > 9.0 g/dL
   * Albumin > 2.7 gm/dL
   * Total bilirubin < 2 mg/dl (Mildly elevated total bilirubin (< 6 mg/dL) is allowed if Gilbert's syndrome is documented)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 5 x ULN
   * Serum creatinine ≤ 1.5 x ULN or creatinine clearance > 50 mL/min (calculated using the Cockcroft-Gault formula)
   * INR/PTT ≤ 1.5 x ULN
   * Alkaline phosphatase limit ≤ 2.5 x ULN
7. At least one measurable (per RECIST 1.1) lesion. Patients who received prior local therapy (e.g., radiofrequency ablation or transarterial chemoembolization, etc.) are eligible provided the target lesion(s) have not been previously treated with local therapy or the target lesion(s) within the field of local therapy have subsequently progressed in accordance with RECIST 1.1.
8. Eastern Cooperative Oncology Group (ECOG) = 0 or 1
9. Negative serum pregnancy test done ≤ 7 days prior to randomization, for females of childbearing potential only.
10. Provide written informed consent.
11. Patients with a prior liver transplant may be included if they have no history of graft rejection within the previous 6 months and stable graft function.

Exclusion Criteria:

1. Prior treatment with regorafenib.
2. Major surgical procedure, open biopsy, or significant traumatic injury ≤28 days prior to randomization.
3. Congestive heart failure > New York Heart Association (NYHA) class 2.
4. Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months) or myocardial infarction less than 6 months prior to randomization.
5. Cardiac arrhythmias requiring anti-arrhythmic therapy. Note: beta blockers or digoxin are permitted.
6. Uncontrolled hypertension. (Systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management).
7. History of or current pheochromocytoma.
8. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism ≤ 6 months prior to randomization.
9. Ongoing infection > grade 2 NCI-CTCAE version 5.0.
10. Patients with seizure disorder requiring medication.
11. Symptomatic metastatic brain or meningeal tumors unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of randomization and is clinically stable with respect to the tumor at the time of randomization.

    NOTE: Patient must not be undergoing acute steroid therapy or taper (chronic steroid therapy is acceptable provided that the dose is stable for one month prior to and following screening radiographic studies).
12. History of organ allograft (including corneal transplant), except prior liver transplant.
13. Hepatic Encephalopathy requiring hospital admission within six (6) months prior to randomization.
14. Ascites requiring paracentesis within four (4) weeks of randomization.
15. Evidence or history of bleeding diathesis or any hemorrhage or bleeding event > CTCAE grade 3 ≤4 weeks prior to randomization.
16. Non-healing wound, ulcer, or bone fracture.
17. Renal failure requiring hemo-or peritoneal dialysis.
18. Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
19. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation.
20. Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
21. Persistent proteinuria of CTC Grade 3 or higher (> 3.5 g/24 hrs, measured by urine protein: creatinine ratio on a random urine sample).
22. Patients unable to swallow oral medications.
23. Any malabsorption conditions that will affect that absorption of regorafenib.
24. Unresolved toxicity greater than CTCAE (version 5.0) Grade 1 attributed to any prior therapy/procedure excluding alopecia and oxaliplatin induced neurotoxicity ≤ Grade 2.
25. Pregnant or nursing women and men or women of childbearing potential who are unwilling to employ adequate contraception because regorafenib is a chemotherapeutic agent that has known genotoxic, mutagenic, and teratogenic effects.

    NOTE: Men and women of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 2 months after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate.
26. Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
27. Immunocompromised patients and patients known to be HIV positive and currently receiving antiretroviral therapy.

NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial. Active infection requiring systemic treatment, known infection with human immunodeficiency virus (HIV), or known acquired immunodeficiency syndrome (AIDS)-related illness 29. Pleural effusion or ascites that causes respiratory compromise (≥ CTCAE version 4.0 Grade 2 dyspnea).

30. Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization) other than study treatment (regorafenib, other agents being investigated in combination with regorafenib).

31. Use of any herbal remedies known to have interference with liver or other major organ functions. Patients must notify the investigator of all herbal remedies used during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 24 months
  The primary objective is to evaluate whether, or not, an 80 mg/day starting dose of regorafenib that escalates weekly by 40 mg until 160 mg/day is non-inferior compared to the FDA approved labeling 160 mg starting dose of regorafenib in terms of Overall Survival in HCC subjects.

SECONDARY OUTCOMES:
Regorafenib treatment cycles | 24 months
  Proportion of patients who complete two cycles of treatment and who intend to initiate Cycle 3 if no progression is noted on the planned 8-week scan
Tumor Progression | 24 months
  Progression-free survival (PFS) per RECIST v1.1 with exploratory analysis of progression-free survival (PFS) per mRECIST where available
Dosing Patterns | 24 months
  Evaluate the dosing schedule of regorafenib treatment, including: cumulative doses received during first and second cycles, duration of treatment (DOT) measured from Cycle 1 Day 1 to the 1 Month Follow-Up 30 days after the last dose of regorafenib, and summary of additional dose patterns or parameters such as the median daily dose for each treatment arm.
EORTC QOL-C30 Quality of Life Measurements | 24 months
  The EORTC QOL-C30 Quality of Life questionnaire contains 30 questions around physical, day-to-day functioning, and side effects experienced measured on a 4 point Likert scale with a response range of "1-not at all," "2-a little bit," "3-quite a bit," and "4-very much." The results between the Arms, particularly for Cycle 1, will be compared.
Optional CD14-16 cell sub-study | 36 months
  An optional sub-study, collect and hold blood samples from 100 subjects for analysis of mononuclear cells (CD14, 15 & 16 cells) and other potential biomarkers at a to-be-determined time point after completion of the study.
FACIT FACT-Hep Quality of Life Measurements | 24 months
  The FACT-Hep Quality of Life questionnaire contains 46 questions around physical, social/family, emotional, day-to-day functioning, and side effects experienced measured on a 5 point Likert scale with a response range of "0-not at all," "1-a little bit," "3-somewhat," "4-quite a bit," and "5-very much." The results between the Arms, particularly for Cycle 1, will be compared..

CONTACTS AND LOCATIONS:
Overall Officials: Catherine T Frenette, MD, Principal Investigator — Scripps MD Anderson Cancer Center; Madappa Kundranda, MD, Principal Investigator — Banner MD Andersen Cancer Center
Locations (9):
- United States (9):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - VA Long Beach Health System, Long Beach, California
  - Tulane University, New Orleans, Louisiana
  - Henry Ford Health Systems, Detroit, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Saint Louis University, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Only aggregated data will be available for review, analysis and reporting.